CLINICAL TRIAL: NCT00537862
Title: Efficacy and Safety of Enteric-coated Mycophenolate Sodium (EC-MPS) in Cyclosporine Microemulsion Based Regimen in de Novo Living Donor Kidney Transplant Recipients ; A Prospective, Open Label, Multi-center Study
Brief Title: Efficacy and Safety of Enteric-coated Mycophenolate Sodium (EC-MPS) in a Cyclosporine Microemulsion Based Regimen in de Novo Living Donor Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERL080AKR02
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplant
Keywords: Kidney Transplant Patients; Immunosuppresion; Enteric-coated mycophenolate sodium

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

SUMMARY:
This study will evaluate the efficacy and safety of enteric-coated mycophenolate sodium (EC-MPS) in a cyclosporine microemulsion based regimen with C2 monitoring in de novo kidney transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* Korean Males and females aged 18 to 65 years.
* Recipients of first, living unrelated or living related non-HLA identical donor kidney
* Transplant, treated with cyclosporine microemulsion (Cs-ME) as primary immunosuppressant.
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to randomization. Effective contraception must be used during the trial and for 6 weeks following discontinuation of the study medication but at least for four months after randomization, even where there has been a history of infertility.

Exclusion Criteria:

* Second or subsequent kidney transplant or multi-organ recipients (e.g. kidney and pancreas) or previous transplant with any other organ.
* Kidneys from cadaveric donors or HLA identical living related donors.
* Patients with any known hypersensitivity to enteric coated Mycophenolate sodium (EC-MPS) or other components of the formulation (e.g. lactose).
* Patients with thrombocytopenia (< 75,000/mm3), with an absolute neutrophil count of <1,500/mm3, and/or leukocytopenia (<4,000/mm3 ), or hemoglobin < 6g/dL .
* Patients who have received any investigational drug within 30 days prior to study entry.
* Patients with a history of malignancy within the last five years, except for successfully excised squamous or basal cell carcinoma of the skin.
* Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception.
* Existence of any surgical or medical condition, other than the current transplant, which in the opinion of the investigator might significantly alter the absorption, distribution, metabolism or excretion of study medication, and/or presence of severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus.
* Patients with clinically significant infection requiring continued therapy.
* Known positive HIV status.
* Positive HBsAg test, or Hepatitis C positive with advanced liver disease or with clinical or pathological diagnosis of cirrhosis.
* Evidence of drug and/or alcohol abuse

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-05; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Efficacy & safety of enteric-coated mycophenolate sodium combined with cyclosporine microemulsion & corticosteroids assessed by overall survival at 6 months, biopsy proven acute rejection, graft loss, adverse events and serious adverse events.

SECONDARY OUTCOMES:
Tolerability of full dose of EC-MPS assessed by dose reduction & treatment discontinuation rates due to adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (4):
- South Korea (4):
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Jeollanam-do
  - Novartis Investigative Site, Seoul